CLINICAL TRIAL: NCT05849480
Title: A Phase I/II Study of CDX-1140, a CD40 Agonist, in Combination With Capecitabine and Oxaliplatin (CAPOX) and Keytruda in Subjects With Biliary Tract Carcinoma (BTC)
Brief Title: A Study of CDX-1140, a CD40 Agonist, in Combination With Capecitabine and Oxaliplatin (CAPOX) and Keytruda in Subjects With Biliary Tract Carcinoma (BTC)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10001548; 001548-C
Record Dates: First submitted 2023-05-08; First posted 2023-05-09 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-22

CONDITIONS: Biliary Cancer; Bile Duct Cancer; Cancer of the Bile Duct
Keywords: Immunotherapy; Pembrolizumab; CAPOX; CDX-1140; CD40 agonist
MeSH Terms: conditions — Biliary Tract Neoplasms; Bile Duct Neoplasms | interventions — Oxaliplatin; Capecitabine; pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase I (Experimental): Keytruda, oxaliplatin, capecitabine and escalating doses of CDX-1140
  Interventions: Drug: oxaliplatin; Drug: capecitabine; Biological: Keytruda; Biological: CDX-1140
- Phase II (Experimental): Keytruda, oxaliplatin, capecitabine and estimated safe dose of CDX-1140
  Interventions: Drug: oxaliplatin; Drug: capecitabine; Biological: Keytruda; Biological: CDX-1140

INTERVENTIONS:
Drug: oxaliplatin — Oxaliplatin (130 mg/m2) will be administered IV on Day 1 of each cycle, every 21 days (up to 6 cycles).
Drug: capecitabine — Capecitabine (750 mg/m2 every 12 hours) will be administered orally with an intermittent schedule: 2 weeks on, 1 week off, of each cycle, every 21 days (up to 6 cycles).
Biological: Keytruda — Pembrolizumab (200 mg) will be given IV on Day 8 of each cycle every 21 days (up to 6 cycles).
Biological: CDX-1140 — CDX-1140 (0.36-1.5 mg/kg; per assigned dose level) will be given IV on Day 8 of each cycle every 21 days (up to 6 cycles).

SUMMARY:
Background:

Biliary tract carcinoma (BTC) is cancer of the slender tubes that carry fluids in the liver. People with advanced BTC have few treatment options, and their survival rates are very low.

Objective:

To test a study drug (CDX-1140) combined 3 other drugs (capecitabine, oxaliplatin, Keytruda) in people with BTC.

Eligibility:

Adults aged 18 years or older with BTC that progressed after treatment and is not eligible for surgery or liver transplant.

Design:

Participants will be screened. They will have a physical exam. They will have blood tests and tests of their heart function. They will have imaging scans. They may need to have a biopsy: A small sample of tissue will be taken from their tumor using a small needle.

Three of the drugs are given through a tube attached to a needle inserted into a vein in the arm (intravenous). The fourth drug is a pill taken by mouth with water.

Participants will be treated in 21-day cycles. They will receive intravenous treatments on day 1 and day 8 of the first 6 cycles. After that, they will receive intravenous treatments only on day 1 of each cycle.

Participants will take the pill twice a day only for the first 2 weeks of each cycle. They will stop taking this drug after 6 cycles.

Imaging scans will be repeated every 9 weeks.

Participants may continue receiving the study treatment for up to 2 years. Follow-up visits, including imaging scans, will continue for 3 more years. These images may be taken at other locations and sent to the researchers.

DETAILED DESCRIPTION:
Background:

Advanced biliary tract carcinoma (BTC) has limited treatment options in the second line setting and a dismal prognosis.

Capecitabine and oxaliplatin (CAPOX) in combination with Keytruda(R) is a tolerable and potentially effective treatment for individuals with refractory advanced BTC.

Programmed cell death protein 1 (PD-1) is an inhibitory receptor that is expressed by all Tcells during activation. It regulates T-cell effector functions during various physiological responses, including acute and chronic infection, cancer and autoimmunity, and immune

homeostasis. Keytruda(R) is a programmed death receptor-1 (PD-1)-blocking antibody indicated for the treatment of different cancers including individuals with hepatocellular carcinoma.

CD40-mediated activation of macrophages and dendritic cells (DC)s in intrahepatic cholangiocarcinoma (iCCA) significantly improves response to anti-PD-1 therapy in preclinical studies. The efficacy of this regimen is enhanced by first-line chemotherapy,

supporting the potential antitumor efficacy of the combination of CD40 agonist antibody (anti-CD40) with anti-PD-1 and chemotherapy.

Objectives:

Phase I: To estimate safe dose of CDX-1140 used in combination with CAPOX, and Keytruda(R)

Phase II:

To evaluate the 6-month progression free survival (PFS) in participants with advanced BTC treated with CDX-1140, CAPOX, and Keytruda(R).

To determine the overall response rate (ORR) defined as complete response (CR) + partial response (PR) according to RECIST 1.1 in participants with advanced BTC.

Eligibility:

Histopathological confirmation of BTC or histopathological confirmation of carcinoma in the setting of clinical and radiological characteristics which, together with the pathology,are highly suggestive of a diagnosis of BTC

Age >=18 years

Evaluable or measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1

Design:

Phase I/II, single-arm, non-randomized trial of Keytruda(R) and CDX-1140 in combination with CAPOX in participants with BTC in the second-line setting.

Initially, 9-12 participants will be enrolled into a Phase I portion of the trial. If safe, we will continue enrollment as planned into Phase II, if not, we will close the protocol.

After estimation of CDX-1140 recommended phase II dose, the first 13 participants enrolled at this dose level of CDX-1140 in Phase I and Phase II will be evaluated for progression. If among these 13 participants, no more than 2 can be progression-free at the 6-months evaluation, then no further participants will be enrolled as soon as this can be determined.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Participants must have histopathological confirmation of BTC or histopathological confirmation of carcinoma in the setting of clinical and radiological characteristics which, together with the pathology, are highly suggestive of a diagnosis of BTC.
  2. The maximum tumor size of any individual tumor or metastasis must be <= 8 cm.
  3. Participants should have progressed on standard of care first line systemic treatment or refused standard treatment.
  4. Participants must have a disease that is not amenable to potentially curative resection or liver transplantation.
  5. Participants must have evaluable or measurable disease per RECIST 1.1
  6. ECOG performance status of 0 to 1
  7. Participants must have adequate organ and marrow function as defined below:

     Absolute neutrophil count

     (ANC) >= 1,000/mcL

     Platelets >= 100,000/mcL

     Total bilirubin <= 2.5 x ULN

     ALT and AST <= 5 x ULN.

     Creatinine OR Measured or calculated creatinine clearance (CrCl) (estimated glomerular filtration rate (eGFR) may also be used in place of CrCl)

     <1.5x institution upper limit of normal OR

     >= 45 mL/min/1.73 m2 for participant with creatinine levels

     >= 1.5 X institutional ULN
  8. Age >=18 years.
  9. Participants must have recovered from any acute toxicity related to prior therapy, including surgery. Toxicity should be <= grade 1. Note: participants with thyroid dysfunction caused by prior therapy including the need for chronic therapy are eligible.
  10. Individuals of child-bearing potential (IOCBP) and individuals able to father a child must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) at the study entry, for the duration of study treatment and up to 4 months after the last dose of the CDX-1140 or Keytruda(R) (all individuals), 9 months (IOCBP), 6 months (individuals able to father a child) after completion of CAPOX therapy whatever comes later
  11. Nursing participants must be willing to discontinue nursing from study treatment initiation through 4 months after study treatment discontinuation.
  12. HBV-infected participants must be on antivirals and have HBV DNA <100 IU/mL. HCV-infected participants can be enrolled if HCV RNA level is undetectable.
  13. Participants must be able to understand and willing to sign a written informed consent document.

EXCLUSION CRITERIA:

1. Participants who have had standard-of-care anti-cancer therapy or therapy with investigational agents (e.g., chemotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, or other investigation agents) or large field radiotherapy within 4 weeks prior to treatment initiation.
2. Prior therapy with anti- CD40.
3. Receiving of live vaccines within 30 days prior to the treatment initiation. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever, rabies, Bacillus Calmette-Guerin, and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist(R)) are live attenuated vaccines and are not allowed.
4. Major surgery within 4 weeks prior to treatment initiation.
5. Active central nervous system metastases and/or carcinomatous meningitis.
6. HIV-infected participants.
7. History of (non-infectious) pneumonitis or current pneumonitis.
8. History of allergic reactions attributed to compounds of similar chemical or biologic composition to study drugs or other agents used in study, such as nivolumab, dacetuzumab, APX005M, ADC-1013.
9. Prior invasive malignancies within the past 3 years prior to treatment initiation (with the exception of non-melanoma skin cancers, non-invasive bladder cancer, or localized prostate cancer for whom systemic therapy is not required).
10. Any medical condition that requires chronic systemic steroid therapy, or any other form of immunosuppressive medication (inhaled and topical steroids are permitted).
11. History of chronic autoimmune disease (e.g., Addison's disease, multiple sclerosis, Graves' disease, Hashimoto's thyroiditis, rheumatoid arthritis, hypophysitis, systemic lupus erythematosus, Wegener's granulomatosis, sarcoidosis syndrome, etc.) or other connective tissue diseases with the symptomatic disease within the 3 years of initiation of study treatment. Note: Active vitiligo or a history of vitiligo will not be a basis for exclusion.
12. Fridericia's corrected QT interval (QTcF) >= 480 msec or other factors that increase the risk of QT prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome.
13. Participants who were not able to tolerate prior immune checkpoint inhibitor therapy.
14. Uncontrolled intercurrent illness or psychiatric illness/social situations that would limit compliance with study requirements.
15. Pregnancy.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2040-06-01 (Estimated); Study Completion 2042-06-01 (Estimated)

PRIMARY OUTCOMES:
Phase I: Safe dose of CDX-1140 in combination with CAPOX and Keytruda(R) | 35 days
  Estimation of safe dose will be determined based on number of dose limiting toxicities (DLTs) experienced.
Phase II: 6-month progression free survival (PFS) probability | Study start - 6 months after start of study drug
  6-month PFS probability will be calculated using the Kaplan-Meier method.
Phase II: Overall response rate (ORR) | Study start until disease progression or 5 years after initiation of study therapy, whichever occurs first.
  The fraction of participants who experience a response (PR + CR) evaluated every 9 (+/- 4) weeks. Results will be reported along with 80% and 95% two-sided confidence intervals.

SECONDARY OUTCOMES:
Safety of CDX-1140, CAPOX and Keytruda(R) in participants with advanced BTC as determined by toxicities experienced | Day 1 of Cycle 1 through 90 days after the study agents were last administered
  Any adverse events/toxicities identified will be reported by type and grade.
5-year overall survival | Study start - 5 years
  Participants will be assessed for survival at study visits while on study therapy and annually thereafter.

CONTACTS AND LOCATIONS:
Overall Officials: Tim F Greten, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP. All collected IPD will be shared with collaborators under the terms of collaborative agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001548-C.html